CLINICAL TRIAL: NCT02441387
Title: Clinical Characteristics and Structural Changes in Magnetic Resonance Imaging: Importance for the Outcome of Late Life Depression
Brief Title: Predictors of the Outcome of Late Life Depression
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Other Study IDs: PREDLLD10446
Record Dates: First submitted 2014-07-10; First posted 2015-05-12 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Major Depression
Keywords: depression; elderly; remission; treatment response; predictors of response; cognitive decline; structural neuroimage; genetic polymorphism; psychoeducation
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Cognitive Dysfunction | interventions — Antidepressive Agents; Sertraline; Escitalopram; Venlafaxine Hydrochloride; Mirtazapine; Therapeutics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — Peripheral venous blood (10mL) will be collected from participants, venocubital puncture into tubes with anticoagulant ethylenediamine tetraacetic acid (EDTA). After collection, the tubes will be properly stored at 4 ° C until the time of extraction. The genomic deoxyribonucleic acid (DNA) will be extracted using a salting out technique (Miller et al. 1988). After DNA extraction, the achieved concentration will be measured by reading the Gene Quant spectrophotometer (Pharmacia Biotech).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Antidepressant treatment: According to their previous treatment history and clinical presentation, patients may take:
  Sertraline 50-250mg/day for 1 year or Escitalopram 10-20mg/day for 1 year or Mirtazapine 15-45mg/day for 1 year or Venlafaxine 37,5-300mg/day for 1 year or Lithium 300-900mg/day for 1 year.
  Interventions: Drug: Antidepressant; Other: Treatment as usual (only pharmacological treatment).
- Antidepressant treatment & Psychoeducation intervention: Antidepressant treatment and psych education program (10 weekly sessions).
  Interventions: Drug: Antidepressant; Other: Psychoeducation

INTERVENTIONS:
Drug: Antidepressant — Sertraline 50-250mg/day for 1 year or Escitalopram 10-20mg/day for 1 year or Mirtazapine 15-45mg/day for 1 year or Venlafaxine 37,5-300mg/day for 1 year or Lithium 300-900mg/day for 1 year.
  Other Names: zoloft, lexapro, efexor, remeron, carbolithium
Other: Psychoeducation — Patients who are in the antidepressant treatment group and does not reach remission (MADRS score <or =8) until visit 4 will be invited to be part of a psychoeducation program. If the patient accepts the psychoeducation intervention, he will be randomized to psychoeducation (pharmacological treatment plus psychoeducation) or treatment as usual (only pharmacological treatment). The psychoeducation program consists of 10 individual sessions, conducted by a trained psychologist who will explain the main concepts of depression and its symptoms, the importance of adhering to treatment, the main side effects of pharmacological treatment, and how to cope with daily difficulties.
  Groups: Antidepressant treatment & Psychoeducation intervention
Other: Treatment as usual (only pharmacological treatment). — Patients who are in the antidepressant treatment group and does not reach remission (MADRS score <or =8) until visit 4 will be invited to be part of a psychoeducation program. If the patient accepts the psychoeducation intervention, he will be randomized to psychoeducation (pharmacological treatment plus psychoeducation) or treatment as usual (only pharmacological treatment).
  Groups: Antidepressant treatment

SUMMARY:
Predictors of response to pharmacological treatment of major depressive disorder will be investigated. One hundred and twenty patients will be included in a naturalistic clinical trial. Psychopathology, personality traits, cognitive performance, brain structural changes and genetic polymorphisms will be evaluated. Patients will be followed for 18 months with a pharmacological treatment algorithm and will be evaluated monthly until 6th month and every 3 months, up to 18 months. Psychoeducation will be offered to patients who did not remit until 3 months of pharmacological tretment.

DETAILED DESCRIPTION:
The relevance of depression prevention and treatment in older people tend to raise in future years, considering the rapid increase of the elderly population in Brazil and the growing impact of depression (the third cause of global burden of diseases in the world according to the World Health Association 2004 report). The association between structural brain changes and treatment response in patients with late-life depression (LLD) remains an intriguing area of research. Predictors of response to pharmacological treatment of major depressive disorder will be investigated in 120 elderly patients, who will be included in a naturalistic clinical trial, that will evaluate psychopathology, personality traits, cognitive performance, brain structural changes and genetic polymorphisms. Patients will be followed for 18 months with a treatment algorithm for depression and will be evaluated monthly until 6th month and every 3 months, up to 18 months, to assess factors associated to response to treatment.

Patients who are in the antidepressant treatment group and does not reach remission (MADRS score <or =8) until 3 months of pharmacological treatment will be invited to be part of a psychoeducation program. If the patient accepts the psychoeducation intervention, he will be randomized to psychoeducation (pharmacological treatment plus psychoeducation) or treatment as usual (only pharmacological treatment). The psychoeducation program consists of 10 individual weekly sessions, conducted by a trained psychologist who will explain the main concepts of depression and its symptoms, the importance of adhering to treatment, the main side effects of pharmacological treatment, and how to cope with daily difficulties.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old
* Major depression (DSMIV-TR)
* Evaluated with MINI
* Willing to participate.

Exclusion Criteria:

* Less than 60 years old
* Dementia syndrome
* Delirium or other organic mental disorders
* Alcohol/drug dependence
* Anxiety disorders, or other psychiatric disorders, and not willing (or not able) to participate

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are 60 years old or older with Major Depression (DSMIV-TR).
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Montgomery-Asberg Depression Scale (MADRS) below 8 during the initial 12 weeks of the study and remained below 8 until 18 months | 18 months
  The investigators will consider patients remitted when their MADRS scale score decreased below 8 during the initial 12 weeks of the study and remained below 8 until 24 weeks. All patients whose MADRS scores decreased to 8 but rose above 8 during the study or whose MADRS score remained at 8 or above throughout the study were considered not remitted

SECONDARY OUTCOMES:
Change from baseline Clinical Global Impression (CGI) up to 18 months | 18 months
  It will be applied on 1st, 2nd, 3rd, 4th, 5th, 6th, 9th, 12th, 15th, and 18th months of follow-up.
  On the 6th, 12th, and 18th months, the Mini Mental State Examination (MMSE), the Cognitive and self-contained part of the Cambridge Examination for Mental Disorders of the Elderly (CAMCOG)and the Bayer Activities of Daily Living Scale (B-ADL) will be applied.
Change from baseline Hamilton-D Scale (HAM-D) up to 18 months | 18 months
  It will be applied on 1st, 2nd, 3rd, 4th, 5th, 6th, 9th, 12th, 15th, and 18th months of follow-up.
  On the 6th, 12th, and 18th months, MMSE, the CAMCOG and the B-ADL will be applied.
Change from baseline Mini Mental State Examination (MMSE) up to 18 months | 18 months
  It will be applied on 1st, 12th, and 18th months of follow-up. On the 6th, 12th, and 18th months, MMSE, the CAMCOG and the B-ADL will be applied.
Change from baseline Cognitive and self-contained part of the Cambridge Examination for Mental Disorders of the Elderly (CAMCOG) up to 18 months | 18 months
  It will be applied on 1st, 12th, and 18th months of follow-up.
Change from baseline Bayer Activities of Daily Living Scale (B-ADL) up to 18 months | 18 months
  It will be applied on 1st, 12th, and 18th months of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Cassio MC Bottino, phD, Study Director — Old Age Research Group (PROTER), Institute and Department of Psychiatry, Faculty of Medicine; Salma Rose Imanari Ribeiz, phD, Principal Investigator — Old Age Research Group (PROTER), Institute and Department of Psychiatry, Faculty of Medicine
Locations (1):
- University of São Paulo, Faculty of Medicine, Institute and Department of Psychiatry, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided